CLINICAL TRIAL: NCT02202239
Title: Effect of Induction and Maintenance of Anesthesia With Etomidate on Hemodynamics and Oxidative Stress in Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140723
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Hemodynamics; Oxidative Stress; Anesthesia
MeSH Terms: interventions — Midazolam; Etomidate; Propofol; Fentanyl; cisatracurium; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group E (Experimental): Etomidate was used in both induction and maintenance of anesthesia.
  Interventions: Drug: midazolam; Drug: Penehyclidine Hydrochloride Injection; Drug: Etomidate; Drug: Fentanyl; Drug: Cisatracurium Besilate; Drug: Remifentanil; Drug: Sevoflurane
- Group P (Active Comparator): Propofol was used in both induction and maintenance of anesthesia.
  Interventions: Drug: midazolam; Drug: Propofol; Drug: Fentanyl; Drug: Cisatracurium Besilate; Drug: Remifentanil; Drug: Sevoflurane

INTERVENTIONS:
Drug: midazolam — Before induction, midazolam 0.05mg/kg will be injected intravenously.
  Other Names: Li Yue Xi
Drug: Penehyclidine Hydrochloride Injection — Penehyclidine Hydrochloride 0.01mg/kg will be injected intravenously after midazolam is injected.
  Other Names: Chang Tuo Ning
  Arms: Group E
Drug: Etomidate — Induction dose: 0.3 mg/kg. Maintenance dose: 10 μg•kg-1•min-1.
  Other Names: Fu Er Li
  Arms: Group E
Drug: Propofol — Induction dose: 2.0 mg/kg. Maintenance dose: 4 to 6 mg/kg/h.
  Arms: Group P
Drug: Fentanyl — During induction, after injection of etomidate, fentanyl 3 μg/kg will be given intravenously.
Drug: Cisatracurium Besilate — Cisatracurium Besilate 0.14 mg/kg will be used after fentanyl is injected for induction.
  During maintenance, intermittent bolus of cisatracurium will be used for maintain muscle relaxation.
Drug: Remifentanil — Remifentanil will be injected continuously during maintenance of anesthesia.
Drug: Sevoflurane — Sevoflurane of 1% to 2% will be administered via inhalation to keep bispectral index（BIS) between 50 to 55.

SUMMARY:
To explore the effect of induction and maintenance of anesthesia with etomidate on hemodynamics and oxidative stress in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years;
* Diabetic patients preparing for elective surgery;
* Body mass index is between 16 and 30 kg/m2;
* Blood glucose is under 8.3 mmol/kg by oral antidiabetic agents or diet control;
* American Society of Anesthesiology (ASA) Physical Status: Ⅰ or Ⅱ;
* Expected operation duration is between 2 and 8 h;
* Signed informed consent form.

Exclusion Criteria:

* Severe cardiac, cerebral, liver, kidney, lung, endocrine disease or infectious disease;
* Chemotherapy or immunotherapy before the surgery;
* Allergy to trial drug or other contraindication;
* Expected or history of difficult airway;
* Suspected abuse of narcotic analgesia;
* Diseases of neuromuscular system;
* Mentally unstable or has a mental illness;
* Trend of malignant hyperthermia;
* Pregnant or breast-feeding women;
* Attendance of other trial past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | from 10 minutes before induction to 1 h after the surgery
  Mean arterial pressure will be measured 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Central venous pressure | from 10 minutes before induction to 1 h after the surgery
  Central venous pressure will be measured 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Heart rate | from 10 minutes before induction to 1 h after the surgery
  Heart rate will be recorded 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Respiratory rate | from 10 minutes before induction to 1 h after the surgery
  Respiratory rate will be measured 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Oxygen saturation | from 10 minutes before induction to 1 h after the surgery
  Oxygen saturation will be measured 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Blood glucose | from 10 minutes before induction to 1 h after the surgery
  Blood glucose will be measured 10 min before the induction (T0), at intubation (T1), 15 min (T2) after intubation, 1 h after the beginning of the surgery (T3), when the surgery is finished (T4) and 1 h after the end of the surgery (T5).
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Insulin | from 10 minutes before induction to 1 h after the surgery
  Insulin will be measured 10 min before the induction (T0), at intubation (T1), 15 min (T2) after intubation, 1 h after the beginning of the surgery (T3), when the surgery is finished (T4) and 1 h after the end of the surgery (T5).
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.

SECONDARY OUTCOMES:
Super oxide dismutase | from 10 minutes before induction to 1 h after the surgery
  2 ml blood will be collected 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery. The blood will be preserved below -20 ℃ before super oxide dismutase was measured.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Glutathione | from 10 minutes before induction to 1 h after the surgery
  2 ml blood will be collected 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery. The blood will be preserved below -20 ℃ before glutathione was measured.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.
Xanthine oxidase | from 10 minutes before induction to 1 h after the surgery
  2 ml blood will be collected 10 min before the induction (T0), at intubation (T1), 5 min (T2), 15 min (T3) after intubation, 30 min after the beginning of the surgery (T4) and 1 h after the end of the surgery. The blood will be preserved below -20 ℃ before xanthine oxidase dismutase was measured.
  Beginning of the surgery: beginning of skin incision. End of the surgery: skin suture is finished.